Congenital Muscular Dystrophy Ascending Multiple Dose Cohort Study analysing Pharmacokinetics at three dose Levels in Children and Adolescents with Assessment of Safety and Tolerability of Omigapil (CALLISTO)

**Study code: SNT-I-015** 

Phase I study

STATISTICAL ANALYSIS PLAN



| Signatures: | |
|-----------------------------------------------------|------|
| Statistical Analysis Plan was prepared by: | |
| Sofia Männikkö | |
| Study Statistician, Oy 4Pharma Ltd. | Date |
| Statistical Analysis Plan was reviewed/approved by: | |
| Senior Statistician | Date |
| Responsible person from the Sponsor | Date |
| Principal Investigator | Date |



# **Table of Contents**

| 1 <i>A</i> | Abbreviations | 4 |
|------------|------------------------------------------------------------|----|
| 2 I | Introduction | 5 |
| 3 S | Study objectives | 5 |
| 4 I | Design and type of the study | 5 |
| | Sample size considerations | |
| | Analysis sets | |
| 6.1 | | |
| 6.2 | Pharmacokinetic (PK) dataset | 6 |
| 6.3 | Safety dataset | 6 |
| 7 I | Disposition of patients | 6 |
| 8 I | Demographic and other baseline characteristics | 6 |
| 9 ( | Concomitant medication/treatment | 7 |
| 10 | Extent of exposure and compliance | 7 |
| 11 | Pharmacokinetics | 7 |
| 12 | Analysis of safety and tolerability | 7 |
| 12. | | |
| 12. | · | |
| 12. | .3 Other safety variables | 8 |
| 13 | | |
| 13. | $\mathcal{S}$ | |
| 13.<br>13. | | |
| 14 | Deviations from the analyses planned in the study protocol | |
| 15 | Execution of statistical analyses | |
| 16 | Hardware and software | |
| 17 | References | |
| 18 | Appendices | |
| 18. | | |
| 18. | .2 Data listing plan (section 16 in the Study report) | 18 |



#### 1 Abbreviations

AE Adverse Event

AESI Adverse Event of Special Interest
ATC Anatomical Therapeutic Chemical

AUC Area Under the Curve

BMI Body Mass Index

CMD Congenital Muscular Dystrophy

COL6-RD Collagen 6-related dystrophies and myopathies

CRM Continual Reassessment Method

CV Coefficient of Variation EK2 Egen Klassification 2

FEV1 Forced Expiratory Volume during first second of the forced breath

FVC Forced Vital Capacity
HHM Hand held myometry

IFR Inspiratory Flow Reserve

ITT Intention to Treat

JHFT Jebsen Hand Function Test

LAMA2-RD Laminin Alpha 2-related dystrophy

MedDRA Medical Dictionary for Regulatory Activities

MEP Maximum Expiratory Pressure

MFM Motor Function Measure

MIP Maximum Inspiratory Pressure

PCF Peak Cough Flow

PEF Peak Expiratory Flow

PK Pharmacokinetic

PP Per Protocol

PT Preferred Term

PUL Performance Upper Limb

QTcF QT corrected for HR using Fridericia's method

QTcB QT corrected for HR using Bazett's method

SAE Serious Adverse Event SAP Statistical Analysis Plan

SD Standard Deviation SOC System Organ Class



SVC Slow Vital Capacity

TEAE Treatment Emergent Adverse Event

#### 2 Introduction

This Statistical Analysis Plan (SAP) describes the statistical analyses to be conducted for study SNT-I-015, an exploratory phase I study of omigapil. The statistical methods were prospectively planned in the study protocol. This SAP was written during the study conduct and the authors and reviewers of the SAP had access to the study data. This SAP serves as documentation of statistical methods used to derive the endpoints and summarize the study data.

## 3 Study objectives

The study objectives were defined in the study protocol. The primary objective of the study is to establish the pharmacokinetic (PK) profile of omigapil in a range of doses in paediatric and adolescent patients with Congenital Muscular Dystrophy (CMD). The secondary objective is to evaluate the safety and tolerability of omigapil at a range of doses in paediatric and adolescent patients. The tertiary objective is to establish the feasibility of conducting disease-relevant clinical assessments in paediatric and adolescent patients with CMD to aid in the design of future studies.

## 4 Design and type of the study

Study SNT-I-015 is a phase I, open-label, sequential group, ascending oral dose, continual reassessment method (CRM) based model, PK, cohort study with patients randomly assigned to one of the three dose cohorts.

Dose levels were to be defined based on the following rules. Four subjects were to be treated at 0.02 mg/kg (level 1) daily for 12 weeks. In case of no toxicity, dose escalation would occur after every 4 subjects until one or more patients exceed the target AUC<sub>0-24h</sub> range. When exceeding the target range, subsequent dose levels were to be determined from the observed PK. Subsequent patients were to be enrolled in groups of 4 using a CRM- type dose escalation/reduction design with the possibility to interpolate between pre-specified doses (Cheung, 2011). As a result, 4 dose levels of omigapil were used for the randomized groups in the following order, along the study, (0.02 mg/kg, 0.08 mg/kg, 0.04 mg/kg, 0.06 mg/kg).

Patients were stratified by disease type (Laminin Alpha 2-related dystrophy [LAMA2-RD] or Collagen 6-related dystrophies and myopathies [COL6-RD]) and weight and will be similarly represented. One patient was to be assigned from each stratum to each dose-escalating group (cohort), so that the cohorts will have similar representation of disease type and weight, to ensure comparable PK, safety, tolerability and efficacy feasibility assessment data.

## 5 Sample size considerations

A total of 16-20 evaluable patients were planned to be accrued using a CRM-type dose escalation/reduction design with the possibility to interpolate between pre-specified doses. The proposed dosing schedule adapts from a CRM-like algorithm called SAVOR (Cheung, Elkind, 2010) that aims to identify a dose exceeding  $AUC_{0-24h}$  of 33 ng h/ml with a probability of 10% or less. The upper end of the  $AUC_{0-24h}$  of 3-33 ng h/ml was targeted because animal modelling in



CMD-relevant models showed higher efficacy at 1 mg/kg compared to 0.1 mg/kg. By enrolling up to 20 patients, 8-12 subjects were to be assigned to the dose predicted to result in the target  $AUC_{0-24h}$  range (which may be less than the highest dose).

## 6 Analysis sets

# 6.1 Intention-to-treat (ITT) dataset

The ITT dataset will include all enrolled patients who received at least one dose of the study medication and completed at least one post-baseline assessment. The ITT dataset will be used for all analyses related to disease relevant clinical assessments.

### 6.2 Pharmacokinetic (PK) dataset

The PK dataset will include all enrolled patients who received at least one dose of the study medication and completed at least one PK assessment. However, a review of dosing information will be performed by the investigator to consider excluding data in any period or on any day where a subject was judged to have received <80 % or >120% of the scheduled dose of the investigational product. Plasma concentration data will be excluded if concentrations are extremely low relative to other subjects' data; in these cases plasma concentrations will be excluded from all or part of the profile, as appropriate. The PK dataset will be used for all PK analyses.

# 6.3 Safety dataset

The Safety dataset will include all enrolled patients who received at least one dose of study medication. Safety dataset will be used for all the safety analyses.

### 7 Disposition of patients

The number of patients enrolled into the study at screening, the number of patients who failed the screening and the reasons for screening failures will be summarized. The number of patients entering and completing the study will be summarized by dose level and overall. Also, the number of patients who discontinued prematurely, the reasons for premature discontinuations and replacement information will be summarized by dose level and overall. The disposition data will also be presented in a listing format.

### 8 Demographic and other baseline characteristics

All demographic and other baseline characteristics (age, height, weight, body mass index [BMI], gender, ethnicity, race, child-bearing potential, ambulatory status, disease type (LAMA2-RD or COL6-RD), time since CMD diagnosis and use of respiratory aid [Bi-Pap]) will be listed by dose level and summarized with descriptive statistics by dose level. The physical examination findings, medical history and pregnancy test results will be listed by dose level.

Age will be calculated using month of birth and month of baseline (screening) visit as difference in months between baseline and time of birth divided by 12. Height will be estimated from ulna length by using the following formulas (Gauld, 2003, 2004):

Height (male, age <20) = ((4.605\* ulna length [cm]) + (1.308\* age [years]) + 28.003



Height (female, age < 20) = ((4.459\* ulna length [cm]) + (1.315 \* age [years]) + 31.485.

Height and weight will also be presented as percentages of normal growth at the age of the patient (Clinical Growth Charts, U.S. National Center for Health Statistics).

#### 9 Concomitant medication/treatment

Concomitant medication and treatments are coded to WHO drug dictionary version September 2017, and will be listed by dose level, including the Preferred term and ATC classification levels 1 and 4.

# 10 Extent of exposure and compliance

The extent of exposure will be summarized based on the duration of study treatment (days). The duration of study treatment will be listed and summarized with descriptive statistics by dose level.

Compliance will be evaluated as percentage of the daily doses taken (calculated from the estimated volume withdrawn from the bottle and daily dosing volumes) since previous visit. Patients with compliance of 80-120% are considered as compliant. The compliance (as %) will be listed by dose level. In addition, the proportion of compliant patients will be tabulated by dose level.

#### 11 Pharmacokinetics

The analysis of the PK parameters is described in a separate PK Analysis Plan (Appendix 18.3).

## 12 Analysis of safety and tolerability

#### 12.1 Adverse events

All recorded adverse events (AEs) will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA version 20.1). All treatment emergent AEs (TEAEs), i.e. events starting or worsening during study treatment or follow-up will be listed by dose level and tabulated by dose level, system organ class (SOC) and preferred term (PT). Both patient and event counts will be included in the tabulations. In addition, tabulations by severity and causality will be provided. Serious TEAEs (SAEs) and TEAEs leading to discontinuation of study treatment will be summarized as data listings. The AEs occurring during the run-in period will be listed separately.

Adverse events of special interest (AESI) will be summarized by dose level, SOC and PT. Also a listing with PFT information from all visits during the study will be presented together with the AE information for subjects experiencing AESI. The following preferred term will be considered as AESI: Pulmonary function test decreased.

### 12.2 Laboratory safety variables

All laboratory data will be listed by dose level. In addition, descriptive statistics of routinely measured laboratory safety variables at each visit will be computed. Both the absolute values and changes from baseline will be summarized by dose level. Frequencies of out-of-range values (low, normal or high) and clinically significant values defined by the investigator will be summarized by dose level and visit as shift tables.



## 12.3 Other safety variables

ECG results (Heart rate, PR, QRS, RR, QT, QTcF and QTcB times) will be listed by dose level and summarized with descriptive statistics by dose level using absolute values and changes from baseline to post-baseline pre-dose values. Moreover, the changes within each visit from pre to post-dose will be summarized. The ECG interpretation (Normal, Abnormal but not clinically significant or Abnormal and clinically significant) and abnormal QTcF and QTcB results (values >500 ms or changes of >30 ms and of > 60 ms) will be listed by dose level and summarized by visit, time point and dose level as shift tables. The QTcF and QTcB times will be calculated based on the following formulas:

$$QTcF = QT / RR^{1/3}$$
$$QTcB = QT / RR^{1/2},$$

where RR = 60 / HR.

Vital signs results (ulna length, height based on ulna length, weight, saturation of peripheral oxygen, blood pressure, heart rate, respiratory rate, body temperature, ability to stand, ambulatory status) will be listed by dose level and summarized descriptively by visit, time point and dose level. Absolute values, changes from baseline to post-baseline pre-dose values and within visit changes from pre- to post-dose values will be presented in the summaries.

Liver abdominal ultrasound results (liver span, echogenicity, presence of cysts and tumours, bile duct dilatation, gallbladder filled, presence of stones and portal vein dilatation) will be listed by dose level and summarized descriptively by dose level and visit. For the last visit, information on changes in the ultrasound from baseline will be listed.

### 13 Disease relevant clinical assessments

All disease relevant clinical assessment variables will be summarized as data listings by dose level. In addition, descriptive statistics/ frequency tables will be included when appropriate. Both absolute values and changes from baseline (if feasible) will be presented. The descriptive statistics/ frequency tables will be broken down by visit. Relevant background status (age of the patient, ambulatory status and type of disease) and AUC<sub>0-24h</sub> information from PK analysis of plasma concentrations vs time profiles of omigapil will be included in the listings.

# 13.1 Respiratory function testing (hospital spirometry)

Respiratory function tests will be presented as non-normalized values and as percentages of predicted values for Peak Expiratory Flow (PEF), Forced Vital Capacity (FVC), Forced Expiratory Volume during first second of the forced breath (FEV1), Maximum Expiratory Pressure (MEP) and Maximum Inspiratory Pressure (MIP). The equations presented in table 13.1.1 will be used for calculation of the percent predicted values. For the equations presented by race, the Caucasian equation will be used also for the Asian subjects. Due to loss of ambulation/ loss of ability to stand, the height will be estimated from the ulna length for all subjects. Age and height used in the equations will always be the age at the time of the measurement and calculated using month of birth and month of assessment date as time difference in months divided by 12.



Table 13.1.1 Percent predicted equations for respiratory function tests

| | predicted equations for respiratory function tests |
|---|---|
| Value<br>(Reference) | Formula |
| | <u>Caucasian</u> |
| PEF%p | Male (age < 20 years): PEF/((-0.5962–(0.12357*age)) + (0.013135* (age^2))+((0.00024962*(height^2))*1))/60*100<br>Female (age < 18 years): PEF/((-3.6181+(0.60644*age))-(0.016846* (age^2))+((0.00018623*(height^2))*1))/60*100 |
| (Hankinson, 1999) | <u>Black or African-American</u> |
| | Male (age < 20 years): PEF/((-0.2684–(0.28016*age))+(0.018202*(age^2)) +((0.00027333*(height^2))*1))/60*100 Female (age < 18 years): PEF/((-1.2398+(0.16375*age))+ ((0.00019746*(height^2))*1))/60*100 |
| | <u>Caucasian</u> |
| | Male (age < 20 years): FVC*100/((-0.2584-( 0.20415*age))+(0.010133* (age^2))+((0.00018642*(height^2))*1)) |
| EVC0/p | Female (age < 18 years): FVC*100/((-1.2082+(0.05916*age))<br>+((0.00014815*(height^2))*1)) |
| FVC%p | <u>Black or African American</u> |
| (Hankinson 1999) | Male (age < 20 years): FVC*100/((-0.4971-(0.15497*age))+ (0.007701*(age^2))+((0.00016643*(height^2))*1)) |
| | Female (age < 18 years): FVC*100/((-0.6166-(0.04687*age))+ (0.003602*(age^2))+ (0.00013606*(height^2))*1)) |
| MEP%p (age < 18) | Male: MEP*100/(7.619+(7.806*age)+(0.004*height*weight)) |
| (Domenech-Clar, 2003) | Female: MEP*100/(17.066+(7.220*age)) |
| MIP%p | M-1 MID#100// 27.020 /4.122# \\ /0.002#1 : 1.# : 1.\\ |
| (Domenech-Clar, 2003) | Male: -MIP*100/(-27.020-(4.132*age)-(0.003*height*weight)) Female: -MIP*100/(-33.854-(1.814*age)-(0.004*height*weight)) |
| FEV1%p | <u>Caucasian</u> |
| (Hankinson 1999) | Male (age < 20 years): FEV1*100/((-0.7453-(0.04106*age))+ (0.004477*(age^2))+((0.00014098*(height^2))*1)) |



| Value<br>(Reference) | Formula |
|---|---|
| | Female (age < 18 years): FEV1*100/((-0.8710+(0.06537*age))+ ((0.00011496*(height^2))*1)) |
| | Black or African American |
| | Male (age < 20 years): FEV1*100/((-0.7048-(0.05711*age))+ (0.004316*(age^2))+((0.00013194*(height^2))*1)) |
| | Female (age < 18 years): FEV1*100/((-0.9630+(0.05799*age))+ ((0.00010846*(height^2))*1)) |

The highest respiratory function test value at each visit will be used in the calculations.

Percent predicted values for PCF will be counted by using the 50<sup>th</sup> percentiles by age presented in table 12.1.2 (Bianchi, 2008) with the following formula: PCF%p = PCF\*100/ 50<sup>th</sup> percentile for the age. Age used in defining the percentiles will be the age at the time of the measurement and calculated with precision using month of birth and month of assessment date.



Table 13.1.2 Percentile values of peak cough flows (liters/min) by gender and age (Bianchi 2008)

| Age, yrs | Females | | | | | | |
|----------|---------|------|------|-------|------|------|-----|
| | 5th | 10th | 25th | 50th | 75th | 90th | 95t |
| 4 | 110 | 112 | 124 | 147 | 179 | 202 | 209 |
| 5 | 125 | 132 | 171 | 185 | 219 | 245 | 273 |
| 6 | 161 | 161 | 191 | 230 | 242 | 284 | 31 |
| 7 | 179 | 200 | 228 | 247 | 265 | 302 | 33 |
| 8 | 200 | 219 | 270 | 299 | 321 | 340 | 35 |
| 9 | 270 | 270 | 290 | 311 | 347 | 369 | 36 |
| 10 | 270 | 284 | 299 | 330 | 361 | 380 | 39 |
| 11 | 296 | 299 | 347 | 380 | 399 | 441 | 47 |
| 12 | 305 | 340 | 361 | 399 | 412 | 450 | 45 |
| 13 | 311 | 330 | 361 | 395 | 441 | 508 | 54 |
| 14 | 361 | 372 | 399 | 428 | 478 | 518 | 56 |
| 15 | 344 | 384 | 424 | 469 | 508 | 550 | 59 |
| 16 | 358 | 412 | 428 | 469 | 508 | 550 | 62 |
| 17 | 369 | 416 | 433 | 469 | 513 | 550 | 63 |
| 18 | 399 | 420 | 441 | 488 | 513 | 556 | 63 |
| | | | | Males | | | |
| Age, yrs | 5th | 10th | 25th | 50th | 75th | 90th | 95t |
| 4 | 130 | 132 | 143 | 162 | 194 | 226 | 23 |
| 5 | 138 | 153 | 179 | 194 | 226 | 262 | 27 |
| 6 | 166 | 171 | 204 | 226 | 250 | 279 | 29 |
| 7 | 200 | 211 | 235 | 270 | 299 | 340 | 35 |
| 8 | 215 | 247 | 279 | 299 | 321 | 340 | 34 |
| 9 | 217 | 237 | 293 | 311 | 340 | 372 | 42 |
| 10 | 250 | 260 | 296 | 321 | 351 | 380 | 42 |
| 11 | 290 | 299 | 340 | 369 | 399 | 420 | 44 |
| 12 | 311 | 317 | 334 | 369 | 399 | 450 | 49 |
| 13 | 321 | 337 | 392 | 450 | 518 | 567 | 57 |
| 14 | 380 | 395 | 498 | 608 | 672 | 713 | 75 |
| 15 | 380 | 428 | 534 | 633 | 706 | 788 | 82 |
| | 493 | 518 | 539 | 652 | 713 | 728 | 87 |
| 16 | | | | | 846 | | 94 |
| 16<br>17 | 498 | 545 | 561 | 645 | 840 | 898 | 94 |

Additionally, Slow Vital Capacity (SVC) will be evaluated as non-normalized values and Inspiratory Flow Reserve (IFR) both as a fraction and as absolute based on the following formulas:

IFR, fraction (%) = 
$$(1 - (V'I, max (t)/ V'I, max (FVC)) *100$$

IFR, absolute = 
$$V'I$$
, max (FVC) –  $V'I$ , max (t).

The best values on the CRF, i.e. the lowest V'I, max (t) and the highest V'I, max (FVC) will be used in the calculations.

For all respiratory parameters, information of use of respiratory aid (Bi-Pap) will be given in the data listings.

## 13.2 Respiratory function testing (handheld ASMA-1 device)

PEF and FEV1 will be presented as non-normalized values and as percent predicted (see equations in 12.1.1). Information of use of respiratory aid (Bi-Pap) will be given in the data listings.



# 13.3 Muscle strength and motor function testing

## 13.3.1 Hand-Held Myometry (HHM)

Knee extension, knee flexion, elbow extension and elbow flexion, measured in Newton units will be presented separately for right and left side. Also, total lower limb score and upper limb score as the sum of extension and flexion results, will be summarized. Upper limb results will also be presented by dominant side. Normalized values (as percentage of normal HHM) will be given for both extension and flexion results. For normalization, the HHM results will be scaled by weight (i.e. knee flexion (N)/ weight (kg)). Average normal HHM values scaled by weight presented by Beenakker (2001) will be used as reference for children aged 4-16. For adults the following formulas from NIH, previously presented by Bohannon (1997), for normalization will be used:

| Knee flexors | e flexors No formula for adults |
|---|---|
| Knee extensors<br>(KE) %p, Female | Dominant side: ((KE/ weight)/(465.22-84.7-(4.803*age)<br>+(0.325*(4.4482216*weight))))*100 |
| | Non-dominant side: ((KE/ weight)/(480.7-95-(4.868*age)+(0.31*(4.4482216*weight))))*100 |
| Knee extensors<br>(KE) %p, Male | Dominant side: ((KE/weight)/(465.22-(4.803*age)<br>+(0.325*(4.4482216*weight))))*100 |
| | Non-dominant side: ((KE/weight)/(480.7-(4.868*age)<br>+(0.31*(4.4482216*weight))))*100 |
| Elbow flexion (EF)<br>%p, Female | Dominant side: ((EF/weight)/(188.36-96.5-(0.61*age)<br>+(0.14*(4.4482216*weight))))*100 |
| | Non-dominant side: ((EF/weight)/(188.25-89.2-(0.65*age)+(0.132*(4.4482216*weight))))*100 |
| Elbow flexion (EF)<br>%p, Male | Dominant side: ((EF/weight)/(188.36-(0.61*age)<br>+(0.14*(4.4482216*weight))))*100 |
| | Non-dominant side: ((EF/weight)/(188.25-(0.65*age)<br>+(0.132*(4.4482216*weight))))*100 |
| Elbow extensors (EE) %p, Female | Dominant side: ((EE/weight)/(156.49-73-(1.032*age)<br>+(0.116*(4.4482216*weight))))*100 |
| | Non-dominant side: ((EE/weight)/(150.37-71.5-(1.044*age)+(0.126*(4.4482216*weight))))*100 |
| Elbow extensors | Dominant side: ((EE/weight)/(156.49-(1.032*age) |



| (EE) %p, Male | +(0.116*(4.4482216*weight))))*100 |
|---|---|
| | Non-dominant side: ((EE/weight)/(150.37-(1.044*age)+(0.126*(4.4482216*weight))))*100 |

## 13.3.2 Goniometry

Goniometry results include measurements of knee extension, elbow extension and ankle dorsiflexion, and the results are presented as grades by side (right/left).

## 13.3.3 Myotools

The Myotools results will be presented as grip strength (kg) and as key pinch (kg) for the dominant hand.

#### 13.3.4 Motor function scales

Jebsen Hand Function Test (JHFT) will be presented as a total score (sec) separately for dominant and non-dominant hand. In addition, data from all subtests will be only listed (without descriptive statistics). For Performance Upper Limb (PUL) and North Star Ambulatory Assessment, total scores will be presented. Moviplate test score values will be presented separately for the dominant hand.

Motor Function Measures (MFM32 or MFM20) will be presented both separately for each dimension (D1 Standing and Transfer, D2 Axial and Proximal Motor Function, D3 Distal Motor function) and as a total score, as % of highest possible scores. In MFM32 the highest possible scores by dimension and in total are D1: 39, D2: 36, D3: 21 and Total: 96. In MFM20 the highest possible scores by dimension and in total are D1: 24, D2: 24, D3: 12 and Total: 60.

#### 13.3.5 Timed tests

The walking distance at 1 and 2 minutes will be presented as meters. In case the subject did not complete the test, the distance at the time the test was stopped will be used for the first missing distance value for the calculation of the descriptive statistics. In this case, the time elapsed when the test was stopped will be shown in the listings.

The time to complete the 10-meter run test and the time to stand from supine will be presented as seconds. In case the subject did not complete the test, the time will be set as missing for the calculation of the descriptive statistics.

Both timed tests will be performed only for ambulatory subjects. Other reasons for not performing the test will be summarized in the listings.

#### 13.3.6 Function scales

The total scores of ACTIVLIM and the Egen Klassification 2 (EK2) will be presented. In addition, the distribution of individual scores by question will be tabulated and the individual scores listed.



## 14 Deviations from the analyses planned in the study protocol

Per protocol analysis will not be conducted because the disease relevant clinical assessments are a tertiary objective of the study, there is no primary disease relevant clinical assessment and while a protocol deviation which is relevant for one organ system may not be relevant for another organ system, definition of a per protocol population is not feasible. Instead, relevant deviations potentially affecting the disease relevant clinical assessments will be discussed case by case on an individual patient and assessment level where appropriate.

## 15 Execution of statistical analyses

Statistical analyses will be performed by Oy 4Pharma Ltd and/or Santhera Pharmaceuticals.

#### 16 Hardware and software

Statistical analysis, tables and patient data listings will be performed with SAS® version 9.3 or higher for Windows (SAS Institute Inc., Cary, NC, USA).

### 17 References

Bianchi C, Baiardi P. (2008) Cough peak flows: standard values for children and adolescents. Am J Phys Med Rehabil.87(6):461-7.

Bohannon RW. (1997) Reference values for Extremity Muscle Strength Obtained by Hand-Held Dynamometry From Adults Aged 20 to 70 Years, Arch Phys Med Rehabil Vol 78, January 1997.

Cheung YK. Dose Finding by the Continual Reassessment Method (2011) New York: Chapman & Hall.

Cheung YK, Elkind MS. (2010) Stochastic approximation with virtual observations for dose-finding on discrete levels Biometrika 97(1):109-121.

Clinical Study Protocol, Final Protocol (01-Dec-2017), Santhera Pharmaceuticals.

Domènech-Clar R, López-Andreu JA, Compte-Torrero L, De Diego-Damiá A, Macián-Gisbert V, Perpiñá-Tordera M, et al. (2003) Maximal static respiratory pressures in children and adolescents. Pediatr Pulmonol. 35(2):126-32.

Gauld LM, Kappers J, Carlin JB, Robertson CF. (2003) Prediction of childhood pulmonary function using ulna length. Am J Respir Crit Care Med. 168(7):804-9.

Gauld LM, Kappers J, Carlin JB, Robertson CF. (2004) Height prediction from ulna length. Dev Med Child Neurol. 46(7):475-80.

Hankinson JL, Odencrantz JR, Fedan KB. (1999) Spirometric Reference Values from a Sample of the General U.S. Population. Am J Respir Crit Care Med Vol 159: 179–187.



## 18 Appendices

# 18.1 Table and figure plan (section 14 in the Study report)

# 14.1 Demographic data

| Table 14.1 | 1 1 Dist | position | of subi | iects |
|------------|----------|----------|---------|-------|

Table 14.1.2.1 Demography and baseline characteristics

Table 14.1.3.1 Analysis datasets

Table 14.1.4.1 Medical history

Table 14.1.5.1 Prior medication and treatments

Table 14.1.5.2 Concomitant medication and treatments

Table 14.1.6.1 Physical examination

Table 14.1.7.1 Pregnancy test results

Table 14.1.8.1 Protocol deviations

Table 14.1.9.1 Compliance to study treatment

## 14.2 Safety data

## 14.2.1 Extent of exposure

Table 14.2.1.1 Extent of exposure

14.2.2 Adverse events

Table 14.2.2.1 Summary of all adverse events

Table 14.2.2.2 Treatment emergent adverse events by SOC and PT

Table 14.2.2.3 Treatment emergent adverse events by PT

Table 14.2.2.4 Treatment emergent adverse events by PT and severity

Table 14.2.2.5 Treatment emergent adverse events by PT and causality

Listing 14.2.2.6 Serious treatment emergent adverse events

Listing 14.2.2.7 Treatment emergent adverse events leading to discontinuation of study treatment

Table 14.2.2.8 Treatment emergent adverse events of special interest

Listing 14.2.2.9 Run-in emergent adverse events

14.2.3 Laboratory results

Table 14.2.3.1 Descriptive statistics of laboratory results

Table 14.2.3.2 Shift table for out of reference range laboratory values

Table 14.2.3.3 Shift table for clinically significant values

14.2.4 ECG results



Table 14.2.4.1 Descriptive statistics of heart rate

Table 14.2.4.2 Descriptive statistics of PR

Table 14.2.4.3 Descriptive statistics of QRS

Table 14.2.4.4 Descriptive statistics of RR

Table 14.2.4.5 Descriptive statistics of QT

Table 14.2.4.6.1 Descriptive statistics of QTcF

Table 14.2.4.6.2 Abnormal QTcF values

Table 14.2.4.7.1 Descriptive statistics of QTcB

Table 14.2.4.7.2 Abnormal QTcB values

Table 14.2.4.8 ECG interpretation

14.2.5 Vital signs

Table 14.2.5.1 Descriptive statistics of ulna length, height based on ulna length and weight

Table 14.2.5.2 Descriptive statistics of saturation of peripheral oxygen

Table 14.2.5.3 Descriptive statistics of blood pressure, heart rate, respiratory rate and body temperature

Table 14.2.5.4 Frequency distributions of being able to stand and ambulatory status

14.2.6 Liver abdominal ultrasound results

Table 14.2.6.1 Frequencies for findings in liver abdominal ultrasound results

#### 14.3 Disease relevant clinical assessments

14.3.1 Respiratory function tests

Table 14.3.1.1 Descriptive statistics respiratory function tests

Figure 14.3.1.2 Individual line plots by cohort for respiratory function tests

14.3.2 ASMA-1 results

Table 14.3.2.1 Descriptive statistics of ASMA-1 results

Figure 14.3.2.2 Individual line plots by cohort for ASMA-1 results

14.3.3 Muscle strength and motor function testing

Table 14.3.3.1 Descriptive statistics of Hand-Held Myometry

Table 14.3.3.2 Descriptive statistics of Goniometry results

Table 14.3.3.3 Descriptive statistics of Myogrip results

Table 14.3.3.4 Descriptive statistics of Jebsen Hand Function Test

Table 14.3.3.5 Descriptive statistics of Performance Upper limb assessment

Table 14.3.3.6 Descriptive statistics of North Star Ambulatory Assessment

Table 14.3.3.7 Descriptive statistics of Moviplate test score



Table 14.3.3.8 Descriptive statistics of Motor Function Measure

14.3.4 Timed tests

Table 14.3.4.1 Descriptive statistics of 2 min walking test distances

Table 14.3.4.2 Descriptive statistics of 10 m run test results

14.3.5 Function scores

Table 14.3.5.1 Descriptive statistics of ACTIVLIM results

Table 14.3.5.2 Descriptive statistics of Egen Klassification 2 results



## 18.2 Data listing plan (section 16 in the Study report)

## 16.2.1 Demographic listings

Listing 16.2.1.1 Inclusion criteria

Listing 16.2.1.2 Exclusion criteria

Listing 16.2.1.3 Medical history

Listing 16.2.1.4 Concomitant medication

Listing 16.2.1.5 Informed consent / Demographic data / Reproductive status

Listing 16.2.1.6 Protocol deviations

Listing 16.2.1.7 Visit dates

Listing 16.2.1.8 End of study information

Listing 16.2.1.9 Populations

Listing 18.2.1.10 Physical examination

# 16.2.2 Compliance and/or Drug concentration data

Listing 16.2.2.1 Dispensing of study medication and dosing

Listing 16.2.2.2 Date of first dose of study medication

Listing 16.2.2.3 Collection of medicine and compliance

## 16.2.3 Individual efficacy response data

Listing 16.2.3.1 Office spirometry

Listing 16.2.3.2 ASMA-1

Listing 16.2.3.3 Muscle strength

Listing 16.2.3.4 Motor function

Listing 16.2.3.5 Timed tests

Listing 16.2.3.6 Functional tests

Listing 16.2.3.7 Muscle imaging

### 16.2.4 Safety data listings

Listing 16.2.4.1 Adverse events

Listing 18.2.4.2 Vital signs

Listing 18.2.4.3 ECG

### 16.2.5 Listing of individual laboratory measurements by subject

Listing 16.2.5.1 Lab data listings: Pharmacokinetics

Listing 16.2.5.2 Lab data listings: Haematology

Listing 16.2.5.3 Lab data listings: Biochemistry

Listing 16.2.5.4 Lab data listings: Urine analysis

Listing 16.2.5.5 Lab data listings: Cardiac and urinary biomarkers